CLINICAL TRIAL: NCT07103577
Title: Guided Island Osteoperiosteal Flap Versus Ridge Splitting for Anterior Atrophic Maxillary Augmentation With Implant Placement (a Randomized Controlled Clinical Trial)
Brief Title: Guided Island Osteoperiosteal Flap Versus Ridge Splitting for Anterior Atrophic Maxillary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0840-01/2024
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Maxillary Alveolar Reconstruction; Virtual Surgical Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computer guided island flap (Experimental)
  Interventions: Procedure: Island osteoperiosteal flap
- Computer guided conventional ridge splitting (Active Comparator)
  Interventions: Procedure: Conventional ridge splitting

INTERVENTIONS:
Procedure: Island osteoperiosteal flap — Crestal incision using no. 15 blade on a bard parker no. 3. Two blind lateral vertical ostotomies at about 1.5 to 2 mm from the adjacent tooth roots to preserve subpapillary and root bone coverage. These cuts are to ensure the complete fracture of buccal plate while being attached to the overlying periosteum.
  Arms: Computer guided island flap
Procedure: Conventional ridge splitting — Crestal incision and 2 vertical releasing incisions will be made using a no.15 blade mounted on a Bard Parker no.3. Then, a full mucoperiosteal flap reflection to expose bone.
  Arms: Computer guided conventional ridge splitting

SUMMARY:
Background: After tooth extraction changes of the shape of the alveolar bone follows a predictable pattern, which proves to be challenging in restoring its form and function, especially in the esthetic zone. Autogenous grafts remain the gold standard because of their predictability. The island osteoperiosteal flap (I-flap) is introduced as a modified alveolar split bone grafting technique used to gain width, height and modify the facial or buccal bone plate position.

Aim of the study: This study aims to evaluate in anterior atrophic maxillary ridge augmentation using guided unreflected island osteoperiosteal flap (I-Flap) approach with simultaneous implant placement and interpostional bone grafting in comparison to computer guided ridge splitting method.

ELIGIBILITY:
Inclusion Criteria:

* Patient seeking replacement of a missed maxillary anterior tooth by a delayed dental implant procedure.
* Residual bone height is (8-15) mm and (3-4) mm alveolar bone width.
* Good oral hygiene.

Exclusion Criteria:

* Uncontrolled Diabetes.
* Coagulation disorders.
* Immunological disorders.
* Previous radiation of the head and neck region.
* Abnormal bone physiology.
* Therapy with Bisphosphonates.
* Heavy smokers.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Change in pain scores | 1 day, 3rd day and 1 week
  Pain (by Visual Analogous Scale):
  Score 0 - No pain. Scores 1 to 3 - Mild pain. Scores 3 to 7 - Moderate pain. scores 7 to 10 - severe pain.
Secondary implant stability | 4 months
  implant stability was measured using ostell device
Change in bone level (bone gain) | Baseline and 4 months
  Immediate post-operative CBCT (T1) will be done to measure the alveolar bone gain, to assess the proper implant positioning, and finally to measure the width of the out-fractured buccal plate and the amount of interpositional bone graft.
  Four months postoperatively CBCT (T2) will be done to measure amount of bone gain
Change in bone density | baseline and 4 months
  Bone density at implant body is measured by using computerized tomography values

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salem OAEH, Elmahlawy AS, Saber ME. Evaluation of 3-Dimensional accuracy of guided implant placement using guided osteoperiosteal flap versus guided ridge splitting for atrophic maxillary augmentation (a randomized clinical trial). BMC Oral Health. 2025 Dec 5;25(1):1905. doi: 10.1186/s12903-025-07364-6. PMID 41350657